CLINICAL TRIAL: NCT02092129
Title: Prognostic Value of Pituitary Histopathology and Plasma Hyperprolactinaemia in Predicting the Risk of Glucose Metabolic Disturbances in Patients With Acromegaly.
Brief Title: Pituitary Histopathology and Hyperprolactinaemia and Risk of Glucose Metabolic Disturbances in Acromegaly.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, Chief Physician, Rigshospitalet, Denmark
Other Study IDs: PROL-BG-ACRO
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Acromegaly; Surgery
Keywords: Acromegaly, surgery, histopathology, hyperprolactinaemia,
MeSH Terms: conditions — Acromegaly; Hyperprolactinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acromegaly: Patients with acromegaly who have received surgical treatment

SUMMARY:
Acromegaly is frequently associated with impaired glucose tolerance and diabetes. We hypothesise that pituitary histopathology and plasma hyperprolactinaemia could have prognostic value in predicting the risk of glucose metabolic disturbances in acromegalic patients. The aim of this study is to examine glucose metabolic outcome in acromegalic patients with and without histologically verified prolactin and growth hormone (GH) co-secreting adenomas. The study population include 79 patients who have all undergone surgical treatment for acromegaly.

DETAILED DESCRIPTION:
Acromegaly is frequently associated with impaired glucose tolerance and diabetes. We hypothesise that pituitary histopathology and plasma hyperprolactinaemia could have prognostic value in predicting the risk of glucose metabolic disturbances in acromegalic patients. The aim of this study is to examine glucose metabolic outcome in acromegalic patients with and without histologically verified prolactin and growth hormone (GH) co-secreting adenomas. 79 patients who have all undergone surgical treatment for acromegaly are included. Clinical and biochemical baseline data are collected from medical records. Patients are divided into two groups based on histopathological evaluation of pituitary adenomas;

1. pure GH secreting adenomas or
2. GH and prolactin co-secreting adenomas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly, and treated at the department of Endocrinology, Copenhagen University Hospital, Rigshospitalet, Denmark (tertiary referral hospital), surgical treatment of acromegaly

Exclusion Criteria:

* no surgical treatment performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acromegaly treated with surgery
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate glucose metabolic outcome related to pituitary histopathology and plasma hyperprolactinaemia in patients with acromegaly | one year
  Patients are grouped according to histopathological evaluation of pituitary adenomas
  1. pure GH secreting adenomas or
  2. GH and prolactin co-secreting adenomas.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- National University Hospital, Department of Medical Endocrinology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No